CLINICAL TRIAL: NCT07052643
Title: Exploring Optimal Photographic Parameters for Standardized Facial Aesthetics Analysis
Acronym: OPTIFACE
Status: Active, not recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1325
Record Dates: First submitted 2025-06-16; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Facial Asymmetry; Reconstructive Surgical Procedures; Facial Morphology
Keywords: Facial Aesthetic; Medical Photography; Facial Analysis; Craniofacial Morphology; Image Standardization
MeSH Terms: conditions — Facial Asymmetry | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Image and data collection — Evaluation of the photographs by four independent raters

SUMMARY:
The main objective of this research is to identify the focal length that allows the most accurate and reproducible 2D assessment of facial aesthetics, without introducing significant distortion. Ultimately, this will enable the establishment of a standardized photography protocol for maxillofacial and aesthetic surgery, facilitating harmonized pre- and post-operative assessments and improving communication between healthcare providers and patients.

DETAILED DESCRIPTION:
Facial aesthetics are a central concern in both reconstructive and aesthetic surgery. Photography has become an essential tool for documenting, comparing, and evaluating facial outcomes before and after surgical procedures. However, variations in camera settings-particularly focal length-can significantly influence the perceived proportions of the face, potentially leading to misinterpretation or distortion in aesthetic assessment.

This project seeks to address this issue by developing a standardized photographic protocol for facial aesthetic evaluation. Specifically, it aims to identify the optimal photographic parameters, with a focus on focal length, that produce the most accurate and consistent two-dimensional (2D) representations of the face. It is well known that different focal lengths affect the visual perception of depth and facial proportions, making the subject appear more or less harmonious or attractive depending on the configuration.

To do this, a collection of facial images will be created using different focal length settings, while keeping other shooting conditions constant (subject-camera distance, lighting, background, and subject posture).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18,
* Signed informed consent

Exclusion Criteria:

* Facial anomalies or Wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the study will be individuals aged 18 years or older, with no recent facial injuries or lesions, and who have provided written informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Identify the focal length setting for optimal assessment of facial aesthetics on 2D photographs | Up to 3 months
  Attractiveness score from 1 to 5 (from very unattractive to very attractive, respectively). The images will be evaluated by 4 independent raters (2 experts: facial surgeons, and 2 non-experts) based on the focal length used: 50 mm, 85 mm, 105 mm, 135 mm, and 200 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas JABALLAH-MAGDELEINE, Principal Investigator — Hôpital NOVO
Locations (1):
- Hôpital NOVO - Site Pontoise, Pontoise, France

IPD SHARING:
Plan to Share IPD: No